CLINICAL TRIAL: NCT05372237
Title: Women's Cardiovascular Health Awareness in Lombardy: a Call for Urgent Appraisal Starting From a Population-based Web-survey: "A Call for Women" Project
Brief Title: Women's Cardiovascular Health Awareness in Lombardy
Acronym: CALLforWOMEN
Status: Completed | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Serenella Castelvecchio, MD, FESC, Principal Investigator, IRCCS Policlinico S. Donato
Other Study IDs: 40/INT/2022
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Cardiovascular Diseases
Keywords: cardiovascular diseases; gender; health awareness; web-survey
MeSH Terms: conditions — Cardiovascular Diseases; Coitus

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiovascular diseases are the leading cause of death in the female population, and it disproportionately affects the young, who are often unaware of their risk profile, which includes both classic and relatively unknown elements. The rise in gestation disorders, depression, and eating disorders among young women must be taken into account. This means that greater awareness starting from the younger generations, and more specific research for women are needed to improve prevention and treatment strategies. "A Call for Women" is an observational study divided into multiple "calls." The first is a web-survey that will be launched in the Lombardy Region with the goal of raising awareness about women's cardiovascular health.

Link for the web-survey [Anticipated]: https://it.surveymonkey.com/r/CallforWomen

DETAILED DESCRIPTION:
[Background] Despite dramatic improvements in the prevention, diagnosis, and treatment of cardiovascular diseases (CVD) in women, CVD continues to be the leading cause of death in women in every major developed country and most emerging economies (1-2). The increasing awareness of sex- (because of the biological factors) and gender differences (those affected by broader social, environmental, and community factors) has stimulated action plans around the world to improve care for women. In the United States, different programs have been launched to promote education among women, including Go Red for Women by the American Heart Association, the Heart Truth by the National Heart, Lung, and Blood Institute, and Make the Call, Don't Miss a Beat by the US Department of Health and Human Services. In doing so, since 1997, the AHA has conducted numerous surveys among US women, proving an increase in awareness of heart disease as the leading cause of death between 1997 and 2012 (from 30% to 56%), especially among younger women (25-34 years of age)(3). Surprisingly, an opposite trend was recently reported. The last released study on behalf of the AHA showed a significant decline in women awareness between 2009 and 2019 (from 65% to 44%), particular in among Hispanic and non-Hispanic Black women and in younger women (in whom primary prevention may be most effective!), calling for an urgent effort to reverse this trend (4). In Europe, such initiatives are scarce, not well organized, with focused plans on a national basis, without adequate dissemination within the scientific community (5). Previous web-based studies have found that around 7% of women (an average number from many ethnic and demographic groups) are aware that heart disease is a real health concern (6). The Italian National Health Service carries out three screening programs for the prevention of tumors, two of which are typically female, breast and cervix, and the third dedicated to both sexes, colorectal. Screening for CVD risk factors is less common in general and in particular among women, without attention for young women and minorities, and most important, has no effect on lowering CVD morbidity and mortality (WHO Health Evidence Network - HEN - synthesis report 7, 2021) Awareness of adverse health conditions, including heart disease, or knowledge of risk factors is the first step in promoting prevention aimed to reduce mortality and morbidity, promoting individual and collective health and well-being. Unfortunately, still today, it is widely believed that cardiovascular diseases concern mainly men, and the great majority of women have a very low perception of the bad outcome caused by these pathologies (7). Furthermore, alongside traditional risk factors, such as high blood pressure, hypercholesterolemia, diabetes, smoking, and overweight, emerging, unrecognized risk factors should be taken into account, including pregnancy-related complications, sedentariness, early menopause, and depression, while potential relationships between eating disorders, lifestyles, chronic inflammatory bowel disease or autoimmune disorders, including celiac disease, and cross complications (e.g., osteopenia and osteoporosis) still deserve to be explored. Surprisingly, the latest released 2021 ESC Guidelines on cardiovascular disease prevention in clinical practice (7) do not recommend systematic CVD risk assessment in women <50 years of age with no known CV risk factors (class III, Level of evidence C), omitting any consideration on potential, emerging risk factors. Indeed, information on whether female-specific conditions improve risk classification is considered a gap in the available evidence. Increasing women's understanding of CVD risk factors and enhancing opportunities to screen women across the lifespan is critical in this scenario with the ultimate goal to better identify women at risk and to improve outcomes. Thus, the first step is to assess the awareness of cardiovascular health and risk factors in a large cohort of women across different social, economic, cultural and health environments.

[Methods] Descriptive observational study, collecting data using a population-based web-survey.

[Study design] Descriptive observational cross-sectional study. The study will be coordinated by a Women Research Group - a multidisciplinary team of women active in the Clinical, Managerial, and Research sectors.

[Data collection] The data will be collected via a population-based web-survey (8-10) created with the SurveyMonkey® software. The collected data will be sent into an electronic data collector, whose output will be saved as an eCRF file in REDCap. The start and end of the data collection are scheduled for April 2022 and April 2023, respectively. Taking into consideration a population of roughly 5 million women in the Lombardy region and an estimated response rate of 80%, the required sample size is calculated in 2182 subjects. More precisely, a sample size of 2182 from a population of 5.000.000 produces a two-sided 80% confidence interval with a precision (half-width) of 0,0070 when the actual proportion is near 0,0700 [from previous web-based studies, roughly 7% of women - an average percentage from several ethnic and demographic groups - were aware regarding CVD (6)]. Consequently, the number of individuals out of the population needed to ask for participation to achieve the required sample size based on the expected response rate is roughly 12.000. The sample size was calculated using the statistical package PASS 2019, v19.0.1.

[Measured variables] All variables will be collected in a self-reporting format. To describe the web-survey-related camp, questions related to socio-demographic profile will be asked, taking into account age, sex, education, and marital status. The proposed item in the population-based web-survey will also face a process of validation: a group of 10/12 health professionals will be asked to express their opinion on the relevance of each item of the questionnaire with regard to the measurement objective of the scale itself. They will express a rating by evaluating each item with a 4-step Likert scale (1 = completely irrelevant; 4 = completely relevant). This approach is useful for content validation and was described by Lawshe (1975) to calculate two quantitative content validation indices (i.e., CVI, CVR). For the face validation (i.e., qualitative validation) three open questions will be asked to the same group of expert clinicians. These questions will be qualitatively analyzed, and any proposals for clarification on the linguistic form of the items will be taken into consideration.

[Statistical analysis] All the data will be checked using the frequency distribution to assess possible missing, errors or outliers. Descriptive statistics will be used to describe the sample characteristics, where categorical data will be presented as frequencies, and continuous data were presented as means ± standard deviation (M±SD) for normally distributed variables, and as median and interquartile range (25°-75° percentile) for continues data non-normally distributed. The study of skewness will be used to preliminary assess the normal distribution of the variables, followed by the Kolmogorov-Smirnov test. Missing data will be managed using a pairwise approach. The sample characteristics will be compared between and within groups and using Pearson's χ2 test for dichotomous variables in the univariate analysis or using The Student's t-test (or one-way ANAOVA when appropriate) for parametric values. Structural equation modellings will test the relationships among the collected health data and to determine whether latent factors might predict the observed variables. Structural equation models will be evaluated considering the interpretation of the following indices of fit: the Satorra-Bentler χ2; the comparative fit index (CFI) (values >0.90 indicated an acceptable fit); the root mean square error of approximation (RMSEA) (values <0.06 indicated an acceptable fit); the weighted root mean square residual (WRMR; values 1.0 indicated an acceptable fit). All data were analyzed using Statistical Package for Social Science version 22 (SPSS, Chicago, IL, USA) and MPLus 8.1, and the level of significance of each test was set at 0.05 and two-tailed.

[Ethical considerations] The study can be described as anonymous because it is impossible to link any particular sample to a person based on the obtained data. Prior to the compilation of the web-survey, the informed consent will be obtained online in the same page. It is not considered necessary to employ a separate written informed permission for this sort of study, according to current legislation (European Regulation 2016/679, Legislative Decree 101/2018), because it would cease to exist the study's confidentiality. On the other hand, it is thought to prioritize properly informing patients with a clear and understandable presentation webpage that explains the survey's purpose before they complete the online questionnaire.

[Data management] All data collected anonymously through the population-based web-survey will be processed in accordance with current legislation (European Regulation 2016/679, Legislative Decree 101/2018), with the GCP and in overall respect of the privacy of the participating subjects, as it will be impossible. for anyone to link any given sample to a subject. The data will be automatically entered into an online binder after each patient completes the questionnaire. Once the collection phase is complete, the binder will be extrapolated into an Excel sheet for analysis purposes. The Excel output will also be deposited in REDCap.

ELIGIBILITY:
Inclusion Criteria:

* Being a woman
* Being over the age of 18
* Residing in the Lombardy region
* Providing informed consent at the start of the population-based web-survey

Exclusion Criteria:

* NOT Being a woman
* NOT Being over the age of 18
* NOT Residing in the Lombardy region
* NOT Providing informed consent at the start of the population-based web-survey

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population-based web-survey will be distributed among women (patients and healthcare providers) at IRCCS Policlinico San Donato but also in the general population via different social, economic and cultural environments also taking advantage of the collaboration of associations already active for women (Fondazione Onda, Soroptimist International, Doppia Difesa - nonprofit organization to protect women victims of violence, etc) or ATS (Health Protection Agency) - Città Metropolitana di Milano.
Sampling Method: Non-Probability Sample
Enrollment: 4969 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2023-11-23 (Actual)

PRIMARY OUTCOMES:
To understand the awareness of CVD risk factors among women in Lombardy using a population-based web-survey | June 2022 (Anticipated) - April 2023 (Anticipated)
  With about 10 million people living in this region, Lombardy forms more than one-sixth of Italy's population, with a reasonable gender employment gap (15% - female employment rate 59.3% vs male employment rate 74.3% / ISTAT data September 2021)

SECONDARY OUTCOMES:
To describe the characteristics of this large cohort of women while measuring their knowledge about health and lifestyle | June 2022 (Anticipated) - April 2023 (Anticipated)
  Increasing women's understanding of CVD risk factors and enhancing opportunities to screen women across the lifespan is critical in this scenario with the ultimate goal to better identify women at risk and to improve outcomes
To describe the healthy/unhealthy behaviors of this large cohort of women | June 2022 (Anticipated) - April 2023 (Anticipated)
  Again, increasing women's understanding of CVD risk factors and enhancing opportunities to screen women across the lifespan is critical in this scenario with the ultimate goal to better identify women at risk and to improve outcomes
To provide epidemiological information to researchers, clinicians and policy-makers about women's CVD | June 2022 (Anticipated) - September 2023 (Anticipated)
  Serving as a catalyst for innovative solutions in screening and teaching campaigns is pivotal for the scientific community

CONTACTS AND LOCATIONS:
Overall Officials: Serenella Castelvecchio, MD, Principal Investigator — IRCCS Policlinico S. Donato
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Milano, Italy

IPD SHARING:
Plan to Share IPD: No
The results from this study will be property of the Promoter and will be used for dissemination through peer-reviewed publications and other forms of scientific communication such as abstracts, oral communications or posters.

REFERENCES:
- [Background] Benjamin EJ, Muntner P, Alonso A, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Das SR, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Jordan LC, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, O'Flaherty M, Pandey A, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Spartano NL, Stokes A, Tirschwell DL, Tsao CW, Turakhia MP, VanWagner LB, Wilkins JT, Wong SS, Virani SS; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2019 Update: A Report From the American Heart Association. Circulation. 2019 Mar 5;139(10):e56-e528. doi: 10.1161/CIR.0000000000000659. No abstract available. PMID 30700139
- [Background] Vaccarino V, Parsons L, Peterson ED, Rogers WJ, Kiefe CI, Canto J. Sex differences in mortality after acute myocardial infarction: changes from 1994 to 2006. Arch Intern Med. 2009 Oct 26;169(19):1767-74. doi: 10.1001/archinternmed.2009.332. PMID 19858434
- [Background] Mosca L, Hammond G, Mochari-Greenberger H, Towfighi A, Albert MA; American Heart Association Cardiovascular Disease and Stroke in Women and Special Populations Committee of the Council on Clinical Cardiology, Council on Epidemiology and Prevention, Council on Cardiovascular Nursing, Council on High Bloo. Fifteen-year trends in awareness of heart disease in women: results of a 2012 American Heart Association national survey. Circulation. 2013 Mar 19;127(11):1254-63, e1-29. doi: 10.1161/CIR.0b013e318287cf2f. Epub 2013 Feb 19. PMID 23429926
- [Background] Cushman M, Shay CM, Howard VJ, Jimenez MC, Lewey J, McSweeney JC, Newby LK, Poudel R, Reynolds HR, Rexrode KM, Sims M, Mosca LJ; American Heart Association. Ten-Year Differences in Women's Awareness Related to Coronary Heart Disease: Results of the 2019 American Heart Association National Survey: A Special Report From the American Heart Association. Circulation. 2021 Feb 16;143(7):e239-e248. doi: 10.1161/CIR.0000000000000907. Epub 2020 Sep 21. PMID 32954796
- [Background] Kouvari M, Souliotis K, Yannakoulia M, Panagiotakos DB. Cardiovascular Diseases in Women: Policies and Practices Around the Globe to Achieve Gender Equity in Cardiac Health. Risk Manag Healthc Policy. 2020 Oct 12;13:2079-2094. doi: 10.2147/RMHP.S264672. eCollection 2020. PMID 33116988
- [Background] Mosca L, Ferris A, Fabunmi R, Robertson RM; American Heart Association. Tracking women's awareness of heart disease: an American Heart Association national study. Circulation. 2004 Feb 10;109(5):573-9. doi: 10.1161/01.CIR.0000115222.69428.C9. Epub 2004 Feb 4. PMID 14761901
- [Background] Visseren FLJ, Mach F, Smulders YM, Carballo D, Koskinas KC, Back M, Benetos A, Biffi A, Boavida JM, Capodanno D, Cosyns B, Crawford C, Davos CH, Desormais I, Di Angelantonio E, Franco OH, Halvorsen S, Hobbs FDR, Hollander M, Jankowska EA, Michal M, Sacco S, Sattar N, Tokgozoglu L, Tonstad S, Tsioufis KP, van Dis I, van Gelder IC, Wanner C, Williams B; ESC National Cardiac Societies; ESC Scientific Document Group. 2021 ESC Guidelines on cardiovascular disease prevention in clinical practice. Eur Heart J. 2021 Sep 7;42(34):3227-3337. doi: 10.1093/eurheartj/ehab484. No abstract available. PMID 34458905
- [Background] Gnambs T, Kaspar K. Disclosure of sensitive behaviors across self-administered survey modes: a meta-analysis. Behav Res Methods. 2015 Dec;47(4):1237-1259. doi: 10.3758/s13428-014-0533-4. PMID 25410404
- [Background] Eysenbach G, Wyatt J. Using the Internet for surveys and health research. J Med Internet Res. 2002 Apr-Nov;4(2):E13. doi: 10.2196/jmir.4.2.e13. PMID 12554560
- [Background] Ball HL. Conducting Online Surveys. J Hum Lact. 2019 Aug;35(3):413-417. doi: 10.1177/0890334419848734. Epub 2019 May 14. PMID 31084575